CLINICAL TRIAL: NCT05603286
Title: Testing an Increased Visit Interval scHeme UsIng Web-based Self-evaluation in Patients With Juvenile Idiopathic Arthritis
Brief Title: Using Self-evaluation to Increase Visit Intervals in Juvenile Idiopathic Arthritis
Acronym: THUIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joeri van Straalen (Other)
Responsible Party: Sponsor-Investigator, Joeri van Straalen, Epidemiologist, coordinating researcher, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NL78722.041.21
Record Dates: First submitted 2022-10-26; First posted 2022-11-02 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: JIA; Self-Evaluation
Keywords: Juvenile idiopathic arthritis; Remote monitoring; E-health; Patient-reported outcomes; Disease activity; Healthcare costs; Non-inferiority trial
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-monitoring arm (Experimental): After inclusion, participants will skip one regular 3-monthly control visit and instead complete an online EQ-5D-Y-5L and JAMAR questionnaire. 5-7 months after inclusion, participants will be followed-up at the hospital and complete a questionnaire about their experiences with home-monitoring.
  Interventions: Procedure: Home-monitoring

INTERVENTIONS:
Procedure: Home-monitoring — Questionnaires for home-monitoring will be send to the participants 11 weeks after the baseline visit via e-mail using Castor EDC and can be completed using a computer, tablet or smartphone. Home-monitoring can be done together with a parent or guardian, if needed.

SUMMARY:
In the THUIS study, JIA patients in clinical remission will skip one 3-monthly hospital control visit and instead monitor their disease activity at home. Outcomes at 6 months will be compared to those from a historical cohort.

DETAILED DESCRIPTION:
Background:

Children with juvenile idiopathic arthritis (JIA) commonly visit their pediatric rheumatologist every 3 months. This costs time and money for the patient, their parents or guardian, the hospital and other stakeholders. Therefore, the THUIS study aims to demonstrate that JIA patients in clinical remission can safely increase their visit interval by home-monitoring disease activity using the EuroQol five-dimensional youth questionnaire with five levels (EQ-5D-Y-5L) and Juvenile Arthritis Multidimensional Assessment Report (JAMAR).

Methods:

JIA patients in remission from the Wilhelmina Children's Hospital in Utrecht, the Netherlands, will skip one 3-monthly control visit and instead complete an online EQ-5D-Y-5L and JAMAR questionnaire at home. The home-monitoring results will be evaluated by a research nurse in consultation with the treating pediatric rheumatologist in order to determine if the patient can safely remain at home or has to be planned in for a short-term control visit at the hospital. Primary and secondary outcomes after 6 months will be compared with a historical cohort of matched JIA patients in order to prove non-inferiority.

ELIGIBILITY:
Inclusion Criteria:

* JIA diagnosis of ≥1 year, all subtypes can participate
* Clinical remission, defined as a cJADAS of ≤3

Exclusion Criteria:

* Insufficient control of the Dutch language
* Not able or willing to use e-mail

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Disease flares | 5-7 months after inclusion.
  The number of disease flares 6 months after baseline visit. A disease flare is defined as a cJADAS score of >3.

SECONDARY OUTCOMES:
Rescheduled visits | Through study completion, an average of 6 months
  The number of rescheduled visits due to presumed disease worsening. Visits can be rescheduled either by the patients themselves or the study team (based on home-monitoring results).
Disease flares at rescheduled visits | Through study completion, an average of 6 months
  The proportion of disease flares observed at rescheduled visits.
Adverse events | Through study completion, an average of 6 months
  The number and type of adverse events reported during follow-up of home-monitoring patients.
Patient satisfaction | 5-7 months after inclusion.
  Patient satisfaction with home-monitoring, measured using a separate 5-item Likert scale questionnaire with higher scores indicating a better outcome.
Reminders | Through study completion, an average of 6 months
  The number of reminders for home-monitoring (via telephone or e-mail) sent to patients.
Failure | Through study completion, an average of 6 months
  The number of patients that fail to home-monitor after two reminders or withdraw from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Joost Swart, MD, PhD, Principal Investigator — Department of Pediatric Immunology and Rheumatology, UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Wilhelmina Children's Hospital, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Study data can be provided by the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication.
Access Criteria: Our study data can be of interest to fellow researchers/clinicians within similar areas interested in increasing visit intervals or home-monitoring in general. Pseudonomized data can be shared with them. The data can also be needed to generate new research questions.

REFERENCES:
- [Background] Doeleman MJH, de Roock S, Buijsse N, Klein M, Bonsel GJ, Seyfert-Margolis V, Swart JF, Wulffraat NM. Monitoring patients with juvenile idiopathic arthritis using health-related quality of life. Pediatr Rheumatol Online J. 2021 Mar 22;19(1):40. doi: 10.1186/s12969-021-00527-z. PMID 33752695